CLINICAL TRIAL: NCT02099929
Title: Coffee and Glucose Metabolism: Clinical, Crossover and Randomized Glucose Disposal Assay Using Stable Isotopes
Brief Title: Effects of Coffee Consumption on Glucose Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Brasilia (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); MRC Human Nutrition Research (Other Government)
Responsible Party: Principal Investigator, Caio Eduardo Gonçalves Reis, Principal Investigator, University of Brasilia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: GliCafé
Record Dates: First submitted 2014-03-26; First posted 2014-03-31 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-03

CONDITIONS: Healthy
Keywords: Coffee; Glucose; Insulin; Diabetes; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Coffee; Sugars; Water

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Coffee with Sugar (Experimental): 300mL of Coffee with 30g of Sugar
  Interventions: Other: Coffee with Sugar
- Coffee without Sugar (Experimental): 300mL of Coffee without Sugar
  Interventions: Other: Coffee without Sugar
- Decaffeinated Coffee without Sugar (Experimental): 300mL of Decaffeinated Coffee without Sugar
  Interventions: Other: Decaffeinated Coffee without Sugar
- Water with Sugar (Sham Comparator): 300mL of Water with 30g of Sugar
  Interventions: Other: Water with Sugar
- Water without Sugar (Sham Comparator): 300mL of Water without Sugar
  Interventions: Other: Water without Sugar

INTERVENTIONS:
Other: Coffee with Sugar — 300mL of Coffee with 30g of Sugar
  Arms: Coffee with Sugar
Other: Coffee without Sugar — 300mL of Coffee without Sugar
  Arms: Coffee without Sugar
Other: Decaffeinated Coffee without Sugar — 300mL of Decaffeinated Coffee without Sugar
  Arms: Decaffeinated Coffee without Sugar
Other: Water with Sugar — 300mL of Water with 30g of Sugar
  Arms: Water with Sugar
Other: Water without Sugar — 300mL of Water without Sugar
  Arms: Water without Sugar

SUMMARY:
Epidemiological studies have shown an inverse association between coffee consumption and risk of type 2 diabetes mellitus (T2DM). However the experimental studies that analysed the mechanisms are limited.

This project aims to assess the effects of coffee consumption on glucose metabolism, using stable isotope tracer (13C-glucose) to explain the possible metabolic mechanisms involved on the reduced risk for T2DM.

DETAILED DESCRIPTION:
This is a crossover randomized clinical trial that has been studying 14 male healthy young adults, who were enrolled five treatments: coffee with sugar, coffee without sugar, decaffeinated coffee without sugar and two controls (water with and without sugar).

The stable isotope minimal model protocol with oral glucose administration (Oral Dose Intravenous Label Experiment - ODILE) was performed. The use of ODILE methodology permits separation of the glucose absorbed and removed from the circulation increasing the accuracy and the effectiveness of glucose uptake and insulin sensitivity (Bluck et al., 2006).

ELIGIBILITY:
Inclusion Criteria:

* Male healthy young adults (18 - 50 years old);
* Body mass index (BMI) between 18.5 - 28.0 kg/m²;
* No weight changes (≥ 5 kg) in the last 3 months;
* Not take any pills/drugs that alter metabolism, appetite and sleep;
* Not have sleep disorders;
* Not have donated blood in the last 3 months;
* Regular breakfast consumption (≥100 kcal ingested up to 2 hours after waking ≥4x/week);
* Being a habitual coffee consumer (≥100mL ≥5x/week).

Exclusion Criteria:

* Diagnosis of anemia, metabolic and heart diseases;
* Previous sudden fainting and convulsions;
* Any drugs and tobacco consumption;
* Consumption of more than 500mg of caffeine / day (5 cups of coffee, tea and cola soft drinks).

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2012-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
ODILE minimal model analysis | -10, 0, 30, 60/0, 15, 30, 45, 47, 49, 51, 53, 55, 57, 59, 61, 65, 70, 75, 80, 85, 90, 100, 115, 135, 165, 195, 225 minutes.
  The stable isotope minimal model protocol with oral glucose administration (Oral Dose Intravenous Label Experiment - ODILE)

SECONDARY OUTCOMES:
Glucose metabolism | -10, 0, 30, 60/0, 15, 30, 45, 47, 49, 51, 53, 55, 57, 59, 61, 65, 70, 75, 80, 85, 90, 100, 115, 135, 165, 195, 225 minutes.
  Glucose and Insulin levels, and Insulin sensitivity indices.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie JC Bluck, PhD, Study Chair — MRC Human Nutrition Research; Teresa HM da Costa, PhD, Study Director — University of Brasilia; Caio EG Reis, MSc, Principal Investigator — University of Brasilia
Locations (1):
- Laboratório de Bioquímica da Nutrição, Núcleo de Nutrição e Medicina Tropical, Universidade de Brasília, Brasília, Federal District, Brazil

REFERENCES:
- [Background] Bluck LJ, Clapperton AT, Coward WA. A stable isotope minimal model protocol with oral glucose administration. Rapid Commun Mass Spectrom. 2006;20(3):493-8. doi: 10.1002/rcm.2326. PMID 16402351